CLINICAL TRIAL: NCT00359788
Title: A Randomized, Double-blind, Parallel Group Trial Comparing 12 Weeks Treatment With Tiotropium 18 mcg Daily to Combivent MDI 2 Actuations Qid in COPD Patients Previously Prescribed Combivent MDI
Brief Title: A Trial Comparing Treatment With Tiotropium Inhalation Capsules to Combivent Inhalation Aerosol in COPD Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 205.325
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Results first posted 2009-11-10 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2013-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Albuterol, Ipratropium Drug Combination; Ipratropium; Albuterol

INTERVENTIONS:
Drug: tiotropium
Drug: Combivent (Ipratropium/Albuterol)

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of 12 weeks treatment with tiotropium HandiHaler 18 micrograms (mcg) daily compared to Combivent Metered Dose Inhaler (MDI) Chlorofluorocarbon Inhalation Aerosol 2 actuations four times a day in Chronic Obstructive Pulmonary Disease (COPD) patients currently prescribed Combivent® MDI.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) Age: greater than or equal to 40 years

* Current or ex-smoker with a >= 10 pack-year smoking history
* Use of Combivent® Metered Dose Inhaler (MDI)for >= 1 month prior to Visit 1

Spirometric criteria (determined at study visits):

* Post-bronchodilator Forced Expiratory Volume in one second (FEV1) <= 70% (Visit 1)
* Pre-bronchodilator FEV1 <= 65% of predicted and FEV1/Forced Vital Capacity (FVC) <= 70% (Visit 2)

Exclusion Criteria:

Clinical history of asthma

* History of thoracotomy with pulmonary resection
* History of Cystic Fibrosis, alpha 1 antitrypsin deficiency or interstitial lung disease
* Daytime use of oxygen therapy for > 1 hour per day or if unable to abstain fr om using oxygen during Pulmonary Function Tests
* Any respiratory tract infection or COPD exacerbation in 6 weeks prior to Visit 1
* Recent history 6 months or less of Myocardial Infarction
* Unstable or life-threatening cardiac arrhythmias
* Hospitalization for Congestive Heart Failure during past year
* Malignancy for which patient is receiving chemo or radiation therapy
* Pregnant or nursing women
* Known hypersensitivity to ipratropium or carrier substances, including related food products such as soybean, peanuts, or lactose
* Use of SPIRIVA® 3 months prior to Visit 1
* Symptomatic of prostatic hypertrophy or bladder neck obstruction
* Known narrow- angle glaucoma
* Participating in a pulmonary rehab program within 4 weeks of Visit 1

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (31):
- United States (31):
  - 205.325.904 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.325.925 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 205.325.909 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 205.325.912 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 205.325.911 Boehringer Ingelheim Investigational Site, Palo Alto, California
  - 205.325.935 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 205.325.903 Boehringer Ingelheim Investigational Site, West Haven, Connecticut
  - 205.325.905 Boehringer Ingelheim Investigational Site, Bay Pines, Florida
  - 205.325.922 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 205.325.907 Boehringer Ingelheim Investigational Site, North Chicago, Illinois
  - 205.325.928 Boehringer Ingelheim Investigational Site, Indiananapolis, Indiana
  - 205.325.923 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 205.325.902 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 205.325.908 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 205.325.920 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 205.325.932 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 205.325.915 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 205.325.914 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 205.325.910 Boehringer Ingelheim Investigational Site, Reno, Nevada
  - 205.325.924 Boehringer Ingelheim Investigational Site, East Orange, New Jersey
  - 205.325.921 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 205.325.917 Boehringer Ingelheim Investigational Site, Buffalo, New York
  - 205.325.926 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.325.901 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 205.325.931 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 205.325.929 Boehringer Ingelheim Investigational Site, Providence, Rhode Island
  - 205.325.936 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 205.325.918 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 205.325.927 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 205.325.919 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 205.325.906 Boehringer Ingelheim Investigational Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Tiotropium: 18 mcg once daily
- Combivent (Ipratropium/Albuterol): 2 actuations 4 times daily
Period: Overall Study
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Started | 173 | 176
Completed | 150 | 159
Not Completed | 23 | 17
Not completed — Adverse Event | 11 | 10
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Protocol Violation | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol) | Total
Number analyzed (Participants) | 173 | 176 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (7.7) | 65.4 (8) | 65.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 33.0
  Male | 153 | 163 | 316.0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 (Forced Expiratory Volume in 1 Second) at 12 Weeks
Description: Trough FEV1 is measured 10 minutes before drug administration
Time Frame: Baseline and 12 Weeks
Population: Participants analyzed belonged to the Full Analysis Set (FAS) and included all patients randomized, treated with study medication and had baseline FEV1 and at least one post-dose trough FEV1.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.081 (0.018) | -0.025 (0.018)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.106, 95% CI 2-sided [0.055 to 0.157]

2. Primary Outcome: Change From Baseline in Average Hourly FEV1 AUC0-6 (Area Under the Curve From Zero to Six Hours) at 12 Weeks
Description: Average hourly FEV1 AUC0-6 minus baseline FEV1
Time Frame: Baseline and 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.187 (0.019) | 0.167 (0.018)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.05 liters; p = 0.0042, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.02, 95% CI [-0.032 to 0.072]

3. Secondary Outcome: Change From Baseline in Trough FEV1 (Forced Expiratory Volume in 1 Second) at 6 Weeks
Description: Trough FEV1 is measured 10 minutes before drug administration
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.11 (0.017) | -0.036 (0.017)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.145, 95% CI [0.098 to 0.193]

4. Secondary Outcome: Change From Baseline in Average Hourly FEV1 AUC0-6 (Area Under the Curve From Zero to Six Hours) on Day 1
Description: Average hourly FEV1 AUC0-6 minus baseline FEV1
Time Frame: Day 1 (after first dose)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.132 (0.012) | 0.211 (0.012)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.08, 95% CI [-0.114 to -0.046]

5. Secondary Outcome: Change From Baseline in Average Hourly FEV1 AUC0-6 (Area Under the Curve From Zero to Six Hours) at Week 6
Description: Average hourly FEV1 AUC0-6 minus baseline FEV1
Time Frame: Baseline and week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.207 (0.019) | 0.153 (0.018)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0447, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.054, 95% CI [0.001 to 0.106]

6. Secondary Outcome: Change From Baseline in Peak FEV1 (Forced Expiratory Volume in 1 Second) on Day 1
Description: Peak FEV1 is defined as the maximum FEV1 observed in the first three hours after dose of study medication
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.232 (0.014) | 0.364 (0.014)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.131, 95% CI [-0.171 to -0.092]

7. Secondary Outcome: Change From Baseline in Peak FEV1 (Forced Expiratory Volume in 1 Second) at Week 6
Description: Peak FEV1 is defined as the maximum FEV1 observed in the first three hours after dose of study medication
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.204 (0.014) | 0.356 (0.013)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.152, 95% CI [-0.19 to -0.113]

8. Secondary Outcome: Change From Baseline in Peak FEV1 (Forced Expiratory Volume in 1 Second) at Week 12
Description: Peak FEV1 is defined as the maximum FEV1 observed in the first three hours after dose of study medication
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.209 (0.015) | 0.342 (0.015)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.133, 95% CI [-0.175 to -0.091]

9. Secondary Outcome: Change From Baseline in Trough FVC (Forced Vital Capacity) at 12 Weeks
Description: Trough FVC is measured 10 minutes before drug administration
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.225 (0.039) | 0.051 (0.038)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0015, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.175, 95% CI [0.067 to 0.283]

10. Secondary Outcome: Change From Baseline in Average Hourly FVC AUC0-6 (Area Under the Curve From Zero to Six Hours) at 12 Weeks
Description: Average hourly FVC AUC0-6 minus baseline FVC
Time Frame: Baseline and 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.443 (0.037) | 0.432 (0.036)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.835, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.011, 95% CI [-0.092 to 0.114]

11. Secondary Outcome: Change From Baseline in Trough FVC (Forced Vital Capacity) at 6 Weeks
Description: Trough FVC is measured 10 minutes before drug administration
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.258 (0.036) | -0.02 (0.035)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.278, 95% CI [0.178 to 0.379]

12. Secondary Outcome: Change From Baseline in Average Hourly FVC AUC0-6 (Area Under the Curve From Zero to Six Hours) on Day 1
Description: Average hourly FVC AUC0-6 minus baseline FVC
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.327 (0.028) | 0.484 (0.028)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.157, 95% CI [-0.236 to -0.078]

13. Secondary Outcome: Change From Baseline in Average Hourly FVC AUC0-6 (Area Under the Curve From Zero to Six Hours) at 6 Weeks
Description: Average hourly FVC AUC0-6 minus baseline FVC
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.464 (0.035) | 0.425 (0.035)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.4386, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.039, 95% CI [-0.059 to 0.137]

14. Secondary Outcome: Change From Baseline in Peak FVC (Forced Vital Capacity) on Day 1
Description: Peak FVC is defined as the maximum FVC observed in the first three hours after dose of study medication
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.542 (0.033) | 0.824 (0.032)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -0.282, 95% CI [-0.374 to -0.191]

15. Secondary Outcome: Change From Baseline in Peak FVC (Forced Vital Capacity) at Week 6
Description: Peak FVC is defined as the maximum FVC observed in the first three hours after dose of study medication
Time Frame: baseline and 6 Weeks (after first dose)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.43 (0.031) | 0.791 (0.031)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.361, 95% CI [-0.449 to -0.274]

16. Secondary Outcome: Change From Baseline in Peak FVC (Forced Vital Capacity) at Week 12
Description: Peak FVC is defined as the maximum FVC observed in the first three hours after dose of study medication
Time Frame: Baseline and 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 0.418 (0.032) | 0.703 (0.032)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.286, 95% CI [-0.375 to -0.196]

17. Secondary Outcome: FEV1 at 15 Minutes on Day 1
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.214 (0.012) | 1.389 (0.011)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.175, 95% CI [-0.207 to -0.142]

18. Secondary Outcome: FEV1 at 30 Minutes on Day 1
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.261 (0.013) | 1.429 (0.013)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.168, 95% CI [-0.205 to -0.131]

19. Secondary Outcome: FEV1 at 1 Hour on Day 1
Time Frame: 1 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.272 (0.014) | 1.455 (0.014)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.182, 95% CI [-0.221 to -0.143]

20. Secondary Outcome: FEV1 at 2 Hours on Day 1
Time Frame: 2 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Least Squares Mean
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Least Squares Mean | 1.293 (0.014) | 1.43 (0.014)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.136, 95% CI [-0.175 to -0.097]

21. Secondary Outcome: FEV1 at 3 Hours on Day 1
Time Frame: 3 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.29 (0.015) | 1.375 (0.014)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.084, 95% CI [-0.125 to -0.044]

22. Secondary Outcome: FEV1 at 4 Hours on Day 1
Time Frame: 4 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.284 (0.015) | 1.319 (0.015)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0997, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.035, 95% CI [-0.076 to 0.007]

23. Secondary Outcome: FEV1 at 6 Hours on Day 1
Time Frame: 6 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.269 (0.016) | 1.233 (0.015)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.101, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.037, 95% CI [-0.007 to 0.08]

24. Secondary Outcome: FEV1 at -10 Minutes at Week 6
Time Frame: 10 minutes before dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.254 (0.017) | 1.108 (0.017)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.145, 95% CI [0.098 to 0.193]

25. Secondary Outcome: FEV1 at 15 Minutes at Week 6
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.3 (0.019) | 1.355 (0.019)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0411, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.055, 95% CI [-0.108 to -0.002]

26. Secondary Outcome: FEV1 at 30 Minutes at Week 6
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.328 (0.02) | 1.388 (0.02)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0354, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.06, 95% CI [-0.116 to -0.004]

27. Secondary Outcome: FEV1 at 1 Hour at Week 6
Time Frame: 1 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.343 (0.021) | 1.405 (0.021)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.041, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.062, 95% CI [-0.121 to -0.003]

28. Secondary Outcome: FEV1 at 2 Hours at Week 6
Time Frame: 2 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.364 (0.021) | 1.382 (0.02)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.5387, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.018, 95% CI [-0.076 to 0.04]

29. Secondary Outcome: FEV1 at 3 Hours at Week 6
Time Frame: 3 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.371 (0.021) | 1.31 (0.02)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0372, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.061, 95% CI [0.004 to 0.118]

30. Secondary Outcome: FEV1 at 4 Hours at Week 6
Time Frame: 4 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.369 (0.02) | 1.247 (0.02)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.121, 95% CI [0.066 to 0.177]

31. Secondary Outcome: FEV1 at 6 Hours at Week 6
Time Frame: 6 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.33 (0.019) | 1.168 (0.019)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.162, 95% CI [0.108 to 0.216]

32. Secondary Outcome: FEV1 at -10 Minutes at Week 12
Time Frame: 10 minutes before dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.225 (0.018) | 1.119 (0.018)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.106, 95% CI [0.055 to 0.157]

33. Secondary Outcome: FEV1 at 15 Minutes at Week 12
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.268 (0.019) | 1.351 (0.019)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0023, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.083, 95% CI [-0.136 to -0.03]

34. Secondary Outcome: FEV1 at 30 Minutes at Week 12
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.306 (0.02) | 1.393 (0.019)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0019, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.087, 95% CI [-0.142 to -0.033]

35. Secondary Outcome: FEV1 at 1 Hour at Week 12
Time Frame: 1 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.327 (0.02) | 1.41 (0.02)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0044, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.083, 95% CI [-0.139 to -0.026]

36. Secondary Outcome: FEV1 at 2 Hours at Week 12
Time Frame: 2 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.353 (0.021) | 1.398 (0.02)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.1182, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.046, 95% CI [-0.103 to 0.012]

37. Secondary Outcome: FEV1 at 3 Hours at Week 12
Time Frame: 3 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.353 (0.021) | 1.333 (0.02)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.4814, ANCOVA — ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.02, 95% CI [-0.037 to 0.078]

38. Secondary Outcome: FEV1 at 4 Hours at Week 12
Time Frame: 4 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.337 (0.02) | 1.263 (0.019)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.008, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.074, 95% CI [0.019 to 0.129]

39. Secondary Outcome: FEV1 at 6 Hours at Week 12
Time Frame: 6 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 1.318 (0.019) | 1.182 (0.019)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.136, 95% CI [0.082 to 0.19]

40. Secondary Outcome: FVC at 15 Minutes on Day 1
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 2.938 (0.036) | 3.308 (0.035)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.37, 95% CI [-0.449 to -0.29]

41. Secondary Outcome: FVC at 30 Minutes on Day 1
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.044 (0.03) | 3.4 (0.03)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.356, 95% CI [-0.44 to -0.272]

42. Secondary Outcome: FVC at 1 Hour on Day 1
Time Frame: 1 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.087 (0.033) | 3.444 (0.033)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.357, 95% CI [-0.451 to -0.264]

43. Secondary Outcome: FVC at 2 Hours on Day 1
Time Frame: 2 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.103 (0.033) | 3.388 (0.032)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.285, 95% CI [-0.376 to -0.194]

44. Secondary Outcome: FVC at 3 Hours on Day 1
Time Frame: 3 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.091 (0.033) | 3.261 (0.032)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0003, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.17, 95% CI [-0.261 to -0.079]

45. Secondary Outcome: FVC at 4 Hours on Day 1
Time Frame: 4 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.087 (0.034) | 3.136 (0.033)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.2992, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.05, 95% CI [-0.143 to 0.044]

46. Secondary Outcome: FVC at 6 Hours on Day 1
Time Frame: 6 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.053 (0.034) | 2.972 (0.034)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0984, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.081, 95% CI [-0.015 to 0.177]

47. Secondary Outcome: FVC at -10 Minutes at Week 6
Time Frame: 10 minutes before dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3 (0.036) | 2.722 (0.035)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.278, 95% CI [0.178 to 0.379]

48. Secondary Outcome: FVC at 15 Minutes at Week 6
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.09 (0.037) | 3.279 (0.036)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0004, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.189, 95% CI [-0.293 to -0.086]

49. Secondary Outcome: FVC at 30 Minutes at Week 6
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.158 (0.039) | 3.362 (0.039)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0003, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.204, 95% CI [-0.314 to -0.095]

50. Secondary Outcome: FVC at 1 Hour at Week 6
Time Frame: 1 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.206 (0.04) | 3.388 (0.039)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.012, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.1832, 95% CI [-0.293 to -0.072]

51. Secondary Outcome: FVC at 2 Hours at Week 6
Time Frame: 2 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.227 (0.039) | 3.338 (0.038)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.044, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.097, 95% CI [-0.219 to 0.003]

52. Secondary Outcome: FVC at 3 Hours at Week 6
Time Frame: 3 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.235 (0.039) | 3.185 (0.038)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.3634, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.05, 95% CI [-0.058 to 0.158]

53. Secondary Outcome: FVC at 4 Hours at Week 6
Time Frame: 4 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.23 (0.039) | 3.068 (0.038)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0032, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.163, 95% CI [0.055 to 0.27]

54. Secondary Outcome: FVC at 6 Hours at Week 6
Time Frame: 6 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.190 (0.037) | 2.914 (0.036)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.275, 95% CI [0.173 to 0.378]

55. Secondary Outcome: FVC at -10 Minutes at Week 12
Time Frame: 10 minutes before dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 2.967 (0.039) | 2.792 (0.038)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0015, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.175, 95% CI [0.067 to 0.283]

56. Secondary Outcome: FVC at 15 Minutes at Week 12
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.069 (0.037) | 3.263 (0.036)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0002, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.193, 95% CI [-0.296 to -0.091]

57. Secondary Outcome: FVC at 30 Minutes at Week 12
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.143 (0.039) | 3.358 (0.038)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.215, 95% CI [-0.323 to -0.108]

58. Secondary Outcome: FVC at 1 Hour at Week 12
Time Frame: 1 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.177 (0.04) | 3.375 (0.039)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0006, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.198, 95% CI [-0.309 to -0.086]

59. Secondary Outcome: FVC at 2 Hours at Week 12
Time Frame: 2 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.231 (0.04) | 3.328 (0.04)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0896, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.097, 95% CI [-0.21 to 0.015]

60. Secondary Outcome: FVC at 3 Hours at Week 12
Time Frame: 3 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.226 (0.04) | 3.218 (0.039)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.8937, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.008, 95% CI [-0.103 to 0.118]

61. Secondary Outcome: FVC at 4 Hours at Week 12
Time Frame: 4 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.199 (0.04) | 3.074 (0.039)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0269, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.125, 95% CI [0.014 to 0.236]

62. Secondary Outcome: FVC at 6 Hours at Week 12
Time Frame: 6 hour
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Liters | 3.155 (0.04) | 2.932 (0.04)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0001, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.223, 95% CI [0.111 to 0.335]

63. Secondary Outcome: Day Time Albuterol Use During Week 1
Description: Puffs of rescue albuterol used during the day in week 1
Time Frame: Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.175 (0.084) | 1.217 (0.082)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.7196, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.042, 95% CI [-0.275 to 0.19]

64. Secondary Outcome: Day Time Albuterol Use During Week 2
Description: Puffs of rescue albuterol used during the day in week 2
Time Frame: Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.24 (0.099) | 1.309 (0.096)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.6189, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.069, 95% CI [-0.343 to 0.205]

65. Secondary Outcome: Day Time Albuterol Use During Week 3
Description: Puffs of rescue albuterol used during the day in week 3
Time Frame: Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.337 (0.104) | 1.41 (0.101)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.6197, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.073, 95% CI [-0.36 to 0.215]

66. Secondary Outcome: Day Time Albuterol Use During Week 4
Description: Puffs of rescue albuterol used during the day in week 4
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.287 (0.107) | 1.399 (0.104)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.4582, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.112, 95% CI [-0.408 to 0.184]

67. Secondary Outcome: Day Time Albuterol Use During Week 5
Description: Puffs of rescue albuterol used during the day in week 5
Time Frame: Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.275 (0.11) | 1.345 (0.107)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.6538, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.07, 95% CI [-0.376 to 0.236]

68. Secondary Outcome: Day Time Albuterol Use During Week 6
Description: Puffs of rescue albuterol used during the day in week 6
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.259 (0.126) | 1.405 (0.123)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.4145, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.145, 95% CI [-0.495 to 0.205]

69. Secondary Outcome: Day Time Albuterol Use During Week 7
Description: Puffs of rescue albuterol used during the day in week 7
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.313 (0.116) | 1.398 (0.114)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.6048, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.085, 95% CI [-0.408 to 0.238]

70. Secondary Outcome: Day Time Albuterol Use During Week 8
Description: Puffs of rescue albuterol used during the day in week 8
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.301 (0.119) | 1.471 (0.117)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.3137, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.17, 95% CI [-0.503 to 0.162]

71. Secondary Outcome: Day Time Albuterol Use During Week 9
Description: Puffs of rescue albuterol used during the day in week 9
Time Frame: Week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.369 (0.12) | 1.43 (0.117)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.7195, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.061, 95% CI [-0.395 to 0.273]

72. Secondary Outcome: Day Time Albuterol Use During Week 10
Description: Puffs of rescue albuterol used during the day in week 10
Time Frame: Week 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.351 (0.116) | 1.394 (0.114)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.7947, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.043, 95% CI [-0.367 to 0.282]

73. Secondary Outcome: Day Time Albuterol Use During Week 11
Description: Puffs of rescue albuterol used during the day in week 11
Time Frame: Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.352 (0.127) | 1.445 (0.124)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.6049, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.093, 95% CI [-0.446 to 0.26]

74. Secondary Outcome: Day Time Albuterol Use During Week 12
Description: Puffs of rescue albuterol used during the day in week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 151 | 158
Puffs per day | 1.361 (0.139) | 1.409 (0.137)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.8109, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.047, 95% CI [-0.437 to 0.342]

75. Secondary Outcome: Night Time Albuterol Use During Week 1
Time Frame: Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.493 (0.259) | 2.966 (0.248)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.1471, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.527, 95% CI [-0.186 to 1.24]

76. Secondary Outcome: Night Time Albuterol Use During Week 2
Description: Puffs of rescue albuterol used during the night in week 2
Time Frame: Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.269 (0.19) | 3.004 (0.182)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.3192, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.265, 95% CI [-0.258 to 0.788]

77. Secondary Outcome: Night Time Albuterol Use During Week 3
Description: Puffs of rescue albuterol used during the night in week 3
Time Frame: Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.282 (0.187) | 2.931 (0.18)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.182, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.351, 95% CI [-0.165 to 0.867]

78. Secondary Outcome: Night Time Albuterol Use During Week 4
Description: Puffs of rescue albuterol used during the night in week 4
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.285 (0.193) | 2.921 (0.184)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.1777, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.363, 95% CI [-0.166 to 0.893]

79. Secondary Outcome: Night Time Albuterol Use During Week 5
Description: Puffs of rescue albuterol used during the night in week 5
Time Frame: Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.152 (0.194) | 2.789 (0.185)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.1805, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.363, 95% CI [-0.169 to 0.895]

80. Secondary Outcome: Night Time Albuterol Use During Week 6
Description: Puffs of rescue albuterol used during the night in week 6
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.178 (0.197) | 2.806 (0.188)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.1777, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.372, 95% CI [-0.17 to 0.913]

81. Secondary Outcome: Night Time Albuterol Use During Week 7
Description: Puffs of rescue albuterol used during the night in week 7
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.156 (0.201) | 2.966 (0.193)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.5725, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.159, 95% CI [-0.395 to 0.714]

82. Secondary Outcome: Night Time Albuterol Use During Week 8
Description: Puffs of rescue albuterol used during the night in week 8
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.104 (0.207) | 2.983 (0.198)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.6765, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.121, 95% CI [-0.449 to 0.69]

83. Secondary Outcome: Night Time Albuterol Use During Week 9
Description: Puffs of rescue albuterol used during the night in week 9
Time Frame: Week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.254 (0.208) | 3.006 (0.198)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.3943, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.247, 95% CI [-0.323 to 0.818]

84. Secondary Outcome: Night Time Albuterol Use During Week 10
Description: Puffs of rescue albuterol used during the night in week 10
Time Frame: Week 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.199 (0.203) | 2.909 (0.196)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.3091, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.291, 95% CI [-0.271 to 0.852]

85. Secondary Outcome: Night Time Albuterol Use During Week 11
Description: Puffs of rescue albuterol used during the night in week 11
Time Frame: Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.224 (0.214) | 2.907 (0.205)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.2911, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.317, 95% CI [-0.273 to 0.907]

86. Secondary Outcome: Night Time Albuterol Use During Week 12
Description: Puffs of rescue albuterol used during the night in week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per night
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 143 | 157
Puffs per night | 3.178 (0.238) | 3.069 (0.229)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.7458, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.108, 95% CI [-0.549 to 0.766]

87. Secondary Outcome: Morning Peak Expiratory Flow Rate (PEFR) at Week 1
Time Frame: Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 205.8 (2.1) | 195.1 (2.059)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0004, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 10.698, 95% CI [4.836 to 16.56]

88. Secondary Outcome: Morning PEFR at Week 2
Description: Weekly means for morning PEFR
Time Frame: Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 206.07 (2.594) | 194.81 (2.516)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0023, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 11.257, 95% CI [4.055 to 18.458]

89. Secondary Outcome: Morning PEFR at Week 3
Description: Weekly means for morning PEFR
Time Frame: Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 206.61 (2.816) | 193.83 (2.742)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0015, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 12.772, 95% CI [4.942 to 20.602]

90. Secondary Outcome: Morning PEFR at Week 4
Description: Weekly means for morning PEFR
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 206.76 (2.959) | 193.19 (2.88)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0013, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 13.568, 95% CI [5.342 to 21.795]

91. Secondary Outcome: Morning PEFR at Week 5
Description: Weekly means for morning PEFR
Time Frame: Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 205.6 (3.012) | 193.55 (2.932)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.005, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 12.052, 95% CI [3.676 to 20.428]

92. Secondary Outcome: Morning PEFR at Week 6
Description: Weekly means for morning PEFR
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 206.49 (3.236) | 195.38 (3.158)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0159, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 11.107, 95% CI [2.095 to 20.119]

93. Secondary Outcome: Morning PEFR at Week 7
Description: Weekly means for morning PEFR
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 208.72 (3.377) | 197.66 (3.326)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0219, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 11.057, 95% CI [1.613 to 20.501]

94. Secondary Outcome: Morning PEFR at Week 8
Description: Weekly means for morning PEFR
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 208.88 (3.385) | 195.22 (3.315)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0048, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 13.655, 95% CI [4.207 to 23.104]

95. Secondary Outcome: Morning PEFR at Week 9
Description: Weekly means for morning PEFR
Time Frame: Week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 208.97 (3.621) | 194.74 (3.531)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0058, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 14.231, 95% CI [4.153 to 24.31]

96. Secondary Outcome: Morning PEFR at Week 10
Description: Weekly means for morning PEFR
Time Frame: Week 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 204.83 (3.608) | 193.23 (3.568)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0248, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 11.597, 95% CI [1.483 to 21.71]

97. Secondary Outcome: Morning PEFR at Week 11
Description: Weekly means for morning PEFR
Time Frame: Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 206.47 (3.607) | 195.47 (3.542)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0325, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 11.001, 95% CI [0.924 to 21.079]

98. Secondary Outcome: Morning PEFR at Week 12
Description: Weekly means for morning PEFR
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 150 | 157
Liters/minute | 206.52 (4.408) | 192.44 (3.996)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0153, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 14.074, 95% CI [2.726 to 25.422]

99. Secondary Outcome: Evening PEFR at Week 1
Description: Weekly means for evening PEFR
Time Frame: Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 222.89 (2.459) | 222.64 (2.352)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.6105, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -1.755, 95% CI [-8.532 to 5.022]

100. Secondary Outcome: Evening PEFR at Week 2
Description: Weekly means for evening PEFR
Time Frame: Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 221.97 (2.715) | 221.12 (2.596)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.8249, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.842, 95% CI [-6.642 to 8.326]

101. Secondary Outcome: Evening PEFR at Week 3
Description: Weekly means for evening PEFR
Time Frame: Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 221.23 (2.793) | 218.52 (2.681)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.4896, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 2.71, 95% CI [-5.001 to 10.421]

102. Secondary Outcome: Evening PEFR at Week 4
Description: Weekly means for evening PEFR
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 221.96 (2.933) | 215.06 (2.796)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0935, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 6.898, 95% CI [-1.172 to 14.968]

103. Secondary Outcome: Evening PEFR at Week 5
Description: Weekly means for evening PEFR
Time Frame: Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 217.95 (3.125) | 214.53 (2.977)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.4339, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 3.419, 95% CI [-5.17 to 12.007]

104. Secondary Outcome: Evening PEFR at Week 6
Description: Weekly means for evening PEFR
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 218.45 (3.535) | 219.42 (3.382)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.845, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = -0.971, 95% CI [-10.74 to 8.799]

105. Secondary Outcome: Evening PEFR at Week 7
Description: Weekly means for evening PEFR
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 220.98 (3.63) | 220.79 (3.468)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.9696, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.194, 95% CI [-9.811 to 10.199]

106. Secondary Outcome: Evening PEFR at Week 8
Description: Weekly means for evening PEFR
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 223.33 (3.721) | 218.2 (3.553)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.3252, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 5.129, 95% CI [-5.117 to 15.376]

107. Secondary Outcome: Evening PEFR at Week 9
Description: Weekly means for evening PEFR
Time Frame: Week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 221.47 (3.86) | 217.41 (3.674)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.452, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 4.062, 95% CI [-6.558 to 14.683]

108. Secondary Outcome: Evening PEFR at Week 10
Description: Weekly means for evening PEFR
Time Frame: Week 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 220.46 (3.808) | 216.32 (3.649)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.4388, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 4.14, 95% CI [-6.372 to 14.651]

109. Secondary Outcome: Evening PEFR at Week 11
Description: Weekly means for evening PEFR
Time Frame: Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 218.35 (3.91) | 217.17 (3.724)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.8288, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 1.185, 95% CI [-9.595 to 11.964]

110. Secondary Outcome: Evening PEFR at Week 12
Description: Weekly means for evening PEFR
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 142 | 157
Liters/minute | 219.66 (4.371) | 215.46 (4.19)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.4929, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 4.204, 95% CI [-7.857 to 16.264]

111. Secondary Outcome: Patient Global Evaluation
Description: The Patient Global Evaluation reflected the patient's opinion of their overall condition with respect to chronic obstructive pulmonary disease (COPD). The scale responses were: Poor (1,2). Fair (3,4), Good (5,6) and Excellent (7,8)
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Units on a scale | 4.273 (0.081) | 4.069 (0.079)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0754, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.204, 95% CI [-0.021 to 0.429]

112. Secondary Outcome: Patient Global Evaluation
Description: The Patient Global Evaluation reflected the patient's opinion of their overall condition with respect to COPD. The scale responses were: Poor (1,2). Fair (3,4), Good (5,6) and Excellent (7,8).
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Units on a scale | 4.49 (0.1) | 4.239 (0.098)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0765, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.251, 95% CI [-0.027 to 0.528]

113. Secondary Outcome: Physician Global Evaluation
Description: The Physician Global Evaluation reflected the physician's opinion of the patients overall condition with respect to COPD. The scale responses were: Poor (1,2). Fair (3,4), Good (5,6) and Excellent (7,8).
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Units on a scale | 4.867 (0.076) | 4.716 (0.075)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.163, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.151, 95% CI [-0.061 to 0.363]

114. Secondary Outcome: Physician Global Evaluation
Description: as for outcome 113
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Number analyzed (Participants) | 152 | 158
Units on a scale | 5.057 (0.076) | 4.772 (0.074)
Statistical Analysis 1: Comparison: Tiotropium vs Combivent (Ipratropium/Albuterol); Test type: Superiority or Other; p = 0.0085, ANCOVA; ANCOVA model with terms for treatment and center as fixed effects and baseline as a covariate; Mean Difference (Final Values) = 0.285, 95% CI [0.073 to 0.496]

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug adminsitration
Arm/Group | Tiotropium | Combivent (Ipratropium/Albuterol)
Serious Adverse Events (participants affected / at risk) | 11/173 | 12/176
Other Adverse Events (participants affected / at risk) | 11/173 | 9/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium (N=173) | Combivent (Ipratropium/Albuterol) (N=176)
Atrial Flutter (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Gastroesophageal Reflux disease (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Small intestional obstruction (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 2 | 1
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium (N=173) | Combivent (Ipratropium/Albuterol) (N=176)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.